CLINICAL TRIAL: NCT01658293
Title: Facilitation of Sensory and Motor Recovery by Means of Heat and Cold-water Stimulation on the Paretic Upper Limb of After Stroke: One Year Follow up
Brief Title: Thermal Stimulation for Stroke Patients
Acronym: TSSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Jia-Ching Chen, Department of Rehabilitation Medicine, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB100-25
Record Dates: First submitted 2012-08-01; First posted 2012-08-07 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Stroke; Upper Limb Paresis
Keywords: stroke; follow up; upper limb; rehabilitation
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- thermal stimulation (Experimental): The experimental group receiving heat and cold-water stimulation, 30 minutes a session, five sessions a week for six weeks.
  Interventions: Behavioral: thermal stimulation
- control group (Active Comparator): The control group receiving the similar intensity of ergometer exercise as the experimental group.
  Interventions: Behavioral: control group ergometer exercises

INTERVENTIONS:
Behavioral: thermal stimulation — The heat and cold-water will be added to the thermal group for 30-40minutes a session daily,five sessions a week for six weeks.
  Arms: thermal stimulation
Behavioral: control group ergometer exercises — The control group will be given ergometer exercises with the similar duration as experimental group.
  Arms: control group

SUMMARY:
Sensory and/or motor deficits in upper limb following stroke often have negative impacts on their daily living. Thermal stimulation with hot and cold pack alternatively incorporated into conventional rehabilitation has been reported and proved to be effective for upper limb functional recovery after stroke. However, whether hot- and cold-water stimulation alternatively based on thermal stimulation also has the effect still remains unknown. The aim of present study is to investigate the facilitated effect of hot and cold water stimulation alternatively on upper limb after stroke.

DETAILED DESCRIPTION:
Stroke patients from department of rehabilitation in Tzu Chi general hospital will be recruited and randomized into two groups, one for experimental group and the other for control group. In addition to receiving routine standard rehabilitation for both groups, the experimental group will receive additional hot- and cold-water stimulation alternatively for five times one session, consecutive four sessions a set, one set for 30 minutes a day and five sets a week for six weeks. The control group will be given ergometer exercises with the similar duration as experimental group. Both groups will be evaluated at baseline before TS and every two weeks till six weeks after TS, then at 3, 6 and 12 months for follow-up. A variety of evaluations used in the present study include Semmes-Weinstein monofilaments for sensory functions; Brunnstrom's stage, Fugl-Meyer Assessment Scale and Motricity Index were used for upper limb motor control and strength; Box and block test for hand dexterity. The modified Motor Assessment Scale and Barthel Index are utilized for evaluating general motor functions and daily activity performance, respectively. The modified Ashworth scale is used for change of muscle tone of upper limb.

ELIGIBILITY:
Inclusion Criteria:

* a first-time ischemic or hemorrhagic stroke.
* no severe diabetes or peripheral vascular disease causing sensory deficits.
* no cognition problem and follow directions indicated by therapist during experiment.
* motor deficit of the upper limb under (including) Brunnstrom stage IV, either in the arm or hand.

Exclusion Criteria:

* a cardiac disease or orthopedic problem history,
* medically unstable such as experienced unstable angina, uncontrolled hypertension according to the treating physician, psychological history before stroke.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Scale for stroke upper limb recovery | one year
  The investigators will use the Fugl-Meyer Assessment Scale as the primary outcome measures in this study evaluating at baseline before TS and six weeks after TS, then at 3, 6 and 12 months for follow-up.
motricity index | one year
  The investigators will use the motricity index as the primary outcome measures in this study evaluating at baseline before TS and six weeks after TS, then at 3, 6 and 12 months for follow-up.

SECONDARY OUTCOMES:
Semmes-Weinstein monofilaments for sensory functions | one year
  The investigators selected the Semmes-Weinstein monofilaments for sensory functions as our secondary outcome measures evaluating at baseline before TS and six weeks after TS, then at 3, 6 and 12 months for follow-up.
the modified motor assessment scale | one year
  The investigators used the modified motor assessment scale as the primary outcome measures in this study evaluating at baseline before TS and six weeks after TS, then at 3, 6 and 12 months for follow-up.
Barthel index | one year
  The investigators used the Barthel index as the primary outcome measures in this study evaluating at baseline before TS and six weeks after TS, then at 3, 6 and 12 months for follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Ching Chen, master, Principal Investigator — Tzu Chi Buddhist General Hospital, Hualien, Taiwan
Locations (1):
- Tzu Chi Buddhist General Hospital, Hualien City, Taiwan

REFERENCES:
- [Derived] Chiu YT, Liang CC, Yu Cheng H, Lin CH, Chen JC. Alternating Hot-Cold Water Immersion Facilitates Motor Function Recovery in the Paretic Upper Limb After Stroke: A Pilot Randomized Controlled Trial. Arch Phys Med Rehabil. 2024 Sep;105(9):1642-1648. doi: 10.1016/j.apmr.2024.05.008. Epub 2024 May 10. PMID 38734047